CLINICAL TRIAL: NCT03105414
Title: Etude INCIPAVE: INCidence Des Pneumopathies Acquises Sous Ventilation Chez l'Enfant
Brief Title: INCIPAVE Study: Incidence of Ventilator Acquired Pneumonia in Children
Acronym: INCIPAVE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sylvie Chevret (Other)
Responsible Party: Sponsor-Investigator, Sylvie Chevret, Professor, Assistance Publique - Hôpitaux de Paris
Organization: Assistance Publique - Hôpitaux de Paris (Other)
Other Study IDs: 11-362
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Pneumonia, Ventilator-Associated
Keywords: Mechanical ventilation; Pediatrics; Cross infection; Intensive care; Diagnosis
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Cross Infection; Disease | interventions — Respiration, Artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Mechanical ventilation — Mechanical ventilation

SUMMARY:
Rationale : ventilator associated pneumonia (VAP) has been extensively studied in adults, however, few data exist regarding VAP in the paediatric intensive care population. The Centers for Disease Control (CDC) definition for VAP is regularly updated trying to homogenised practice, and the last version for paediatrics has been published in 2015. According to the latest CDC definition, the investigators aim to study incidence of VAP in different paediatric intensive care units (PICUs), diagnostic methods of identifying VAP, microbiology of VAP, and utilisation of empirical antimicrobial therapy.

Methods and population : a prospective multicentre observational study will be conducted in European PICUs for one year. All patients admitted to PICU aged more than 28 days and < 18 years, mechanically ventilated either by endotracheal or tracheostomy tube are included. Clinical data, ventilation settings, and risk factors for VAP are inserted daily in an electronic database on the internet. The investigators are going to identify patients, who presented one or more episodes of VAP during PICUs stay, analysing onset circumstances, diagnostic methods, bacteria pathogens identified, and antibiotic treatment. VAP incidence will be reported as number of events per 1,000 ventilator-days. Risk factors associated to VAP will be identified by univariate and multivariate analysis.

Results and perspective : the investigators aim to define for the first time the incidence of VAP among European PICUs with a prospective and multicentre study. The identification of risk factors, diagnostic methods, epidemiology, treatment strategies will define the basis to start prevention manoeuvres and improve the clinical strategies for VAP in paediatric intensive care population.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to Pediatric Intensive Care Unit
* Aged more than 28 days and < 18 years
* Mechanically ventilated either by endotracheal or tracheostomy tube

Exclusion Criteria:

-

Ages: 28 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients admitted to Pediatric Intensive Care Unit aged more than 28 days and < 18 years, mechanically ventilated either by endotracheal or tracheostomy tube are included. Clinical data, ventilation settings, and risk factors for VAP are inserted daily in an electronic database on the internet.
Sampling Method: Probability Sample
Enrollment: 2100 (Estimated)
Dates: Start 2017-04-03 (Actual); Primary Completion 2018-05-15 (Estimated); Study Completion 2019-05-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of ventilator acquired pneumonia | Until weaning of ventilator or 1 year
  CDC definition of ventilator acquired pneumonia

SECONDARY OUTCOMES:
Bacteria prevalence of ventilator acquired pneumonia | Until weaning of ventilator or 1 year
prevalence of diagnostic devices used to identify ventilator acquired pneumonia | Until weaning of ventilator or 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Robert Debré Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided